CLINICAL TRIAL: NCT00111982
Title: Multi-Center, Open-Label Trial of Extended Treatment With Liatermin (r-metHuGDNF) Administered by Continuous Intraputaminal (IPu) Infusion to Subjects With Idiopathic Parkinson's Disease Who Have Completed a Previous Trial of Liatermin (Protocol 20020168)
Brief Title: Trial of Extended Treatment With Liatermin (r-metHuGDNF) Administered by Continuous Intraputaminal (IPu)Infusion to Subjects With Idiopathic Parkinson's Disease Who Have Completed a Previous Trial of Liatermin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030160
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Parkinson's Disease
Keywords: bilateral, idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Glial Cell Line-Derived Neurotrophic Factor

ARMS (1):
- Liatermin (Experimental): Bilateral continuous infusion of liatermin for up to 24 months.
  Interventions: Biological: Liatermin

INTERVENTIONS:
Biological: Liatermin — Liatermin

SUMMARY:
The purpose of this study is to determine long-term efficacy of continuous IPu liatermin infusion administered with concomitant standard anti-Parkinsonian therapy.

ELIGIBILITY:
Inclusion Criteria: - Completion of the 20020168 protocol

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2003-12; Primary Completion 2005-11 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Percent change in UPDRS | 24 months

SECONDARY OUTCOMES:
Incidence of treatment emergent and device related adverse events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com